CLINICAL TRIAL: NCT05135377
Title: Canadian Anaphylaxis Network- Predicting Recurrence After Emergency Presentation for Allergic REaction
Acronym: CAN-PREPARE
Status: Active, not recruiting | Type: Observational
Sponsor: Waleed Alqurashi (Other)
Collaborators: Stollery Children's Hospital (Other); Children's Hospital of Western Ontario (Other); The Hospital for Sick Children (Other); Alberta Children's Hospital (Other); McMaster University (Other); CHU Ste-Justine, Montreal (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Waleed Alqurashi, Assistant Professor, MD, MSc, FAAP, FRCPC, Children's Hospital of Eastern Ontario
Organization: Children's Hospital of Eastern Ontario (Other)
Other Study IDs: CTO 3721
Record Dates: First submitted 2021-11-11; First posted 2021-11-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Anaphylaxis
Keywords: Biphasic Anaphylaxis
MeSH Terms: conditions — Anaphylaxis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with Anaphylaxis: Patients under 18 years of age presenting to the Emergency Department (ED) with an allergic reaction that matches diagnostic criteria for anaphylaxis.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Not applicable - observational study

SUMMARY:
BACKGROUND: Anaphylaxis is the most severe form of allergy that rapidly affects multiple body systems and can be deadly. The highest incidence of anaphylaxis is in children and adolescents. In Canada, approximately every 10 minutes there is an Emergency Department (ED) visit for food allergy, and up to 80% of anaphylactic reactions in children are triggered by food. The ambiguity in how physicians manage anaphylaxis adds a huge burden to health care and further contributes to ED crowding. Current Canadian and international treatment guidelines universally recommend that all patients present to the ED for a prolonged period (6-24 hours) of in-hospital monitoring after initial reactions have been treated, to increase detection of biphasic anaphylaxis (BA). BA is a second wave of symptoms after initial resolution. These guidelines are based on poor or little evidence and have unintended negative impacts on patient safety and quality of life. Furthermore, this 'one-size fits all' approach to care leads to wasteful resource utilization that provides low value care.

OBJECTIVE: The main objective of the study is to derive a clinical prediction rule that identifies children with anaphylaxis who are at risk of BA.

METHODS: This prospective multicenter cohort study will enroll 1682 patients from 7 pediatric EDs that are members of the Pediatric Emergency Research Canada (PERC) network. We will enroll patients < 18 years of age presenting to the ED with an allergic reaction that matches the diagnostic criteria of anaphylaxis. Research assistants (RA) present in the ED will screen, obtain consent, and prospectively collect all study data. The Research Assistant or Research Nurse will follow patients during their ED visit and ascertain, in conjunction with the medical team, if the patient developed biphasic anaphylaxis in the ED. A standardized follow-up survey conducted within 2-5 days of ED or hospital discharge will determine if a biphasic reaction occurred following ED disposition. We established an advisory council comprised of end-users and community partners external to the project team to monitor project milestones.

STUDY TEAM: We have established an international multidisciplinary team of experts in pediatrics, emergency medicine, allergy/immunology, research methodology and statistics, and knowledge translation. Our team is supported by the PERC network.

EXPECTED OUTCOME: Providing the best evidence-based, value care at the lowest cost is a moral and ethical imperative. Therefore, in alignment with national and international research priorities, we propose to develop a robust prediction model for BA. This model will address a significant gap in current knowledge and practice, with anticipated benefit for patient care and health system efficiency worldwide. This trial will generate novel, clinically relevant data on optimal ED management of children with anaphylaxis that integrates best value care with patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 18 years of age presenting to the ED with an allergic reaction that matches diagnostic criteria for anaphylaxis as defined by the World Allergy Organization (WAO) in 2019. The 2019 WAO anaphylaxis guidelines clarify the involvement of two organ systems to diagnose anaphylaxis, stating that "although the diagnosis of anaphylaxis usually depends on the involvement of multiple organ systems, anaphylaxis may present as an acute cardiac or respiratory event as the only manifestation of anaphylaxis." Thus, a patient with isolated hypotension, bronchospasm, or upper airway obstruction after exposure to a known or potential trigger will be deemed to have anaphylaxis, even if typical skin features are absent.
* Language proficiency in English or French

Exclusion Criteria:

* Anaphylactic reaction that occurred in the context of a suicidal attempt or intoxication
* Anaphylactic reaction that begins in hospital and managed outside ED (on an inpatient or outpatient unit)
* Patient who is unable to complete the follow-up survey post ED discharge.
* Previous enrollment in the CAN-PREPARE Study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients under the age of 18 who present to the Emergency Department with an allergic reaction that matches diagnostic criteria for anaphylaxis.
Sampling Method: Probability Sample
Enrollment: 1682 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of biphasic anaphylaxis | Up to 5 days post enrollment
  The primary outcome for this prospective cohort study of children who present to ED with anaphylaxis is the development of biphasic anaphylaxis (BA) in the ED or after hospital/ED discharge. As per the published consensus definition in 2019, to be classified as BA, an anaphylactic reaction must meet 3 criteria: 1) initial anaphylactic reaction followed by resolution of all initial manifestations for ≥1 h, with no new symptoms or treatment administered in that time; 2) the second phase of new or recurrent symptoms or signs that meet the consensus definition of anaphylaxis, and 3) the new or recurrent symptoms or signs are not caused by antigen re-exposure. This definition focuses on clinically important or major biphasic reactions. Mild symptoms that involve only the skin (e.g. urticarial rash) without any other systems involvement will be captured and classified as minor biphasic responses. However, these minor responses do not meet our case definition for BA.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Alqurashi, MD, Principal Investigator — Children's Hospital of Eastern Ontario; Amy C Plint, MD, Principal Investigator — Children's Hospital of Eastern Ontario; Marcus S Shaker, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (7):
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - McMaster University, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alqurashi W, Shaker M, Wells GA, Collins GS, Greenhawt M, Curran JA, Zemek R, Schuh S, Ellis A, Gerdts J, Kreviazuk C, Dixon A, Eltorki M, Freedman SB, Gravel J, Poonai N, Worm M, Plint AC. Canadian Anaphylaxis Network-Predicting Recurrence after Emergency Presentation for Allergic REaction (CAN-PREPARE): a prospective, cohort study protocol. BMJ Open. 2022 Oct 31;12(10):e061976. doi: 10.1136/bmjopen-2022-061976. PMID 36316072
- See also: Study Protocol Publication — https://bmjopen.bmj.com/content/12/10/e061976.full